CLINICAL TRIAL: NCT01516385
Title: Detection of Peripheral Blood Biomarkers in Intermediate Phase Spinal Cord Injury: Correlation With Neurological and Functional Outcomes, and Comparison to Other Central and Peripheral Neurological Conditions.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: SHEBA-12-8822-ORK-CTIL
Record Dates: First submitted 2012-01-19; First posted 2012-01-24 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Spinal Cord Injury
Keywords: spinal cord injury; biomarkers; rehabilitation; functional independence; prognosis
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- spinal cord injury
- other neurological conditions

SUMMARY:
This research looks for markers in the blood of people with spinal cord injury that may be a sign of injury severity, or serve as a clue to the degree of recovery. Investigators would also like to compare the marker profile of these patient with that of other neurological conditions such as stroke and Guillain-Barre syndrome.

Patients participating in this trial will be those accepted to neuro-rehabilitation in Sheba medical center, Israel. They will join the trial at their arrival to the ward, no less than 2 week after the beginning of their condition, but no later than 3 months.

Patients will be examined by the research staff three times:

1. At arrival, the patients will be neurologically examined and their functional abilities will be assessed. Blood will be drawn and sent to the lab.
2. At 6 months after the beginning of the neurological condition the same will be repeated: the patients will be neurologically examined and their functional abilities will be assessed, and blood will be drawn and sent to the lab.
3. The final examination will take place 1 year after the beginning of the neurological condition. This time only the neurological and functional abilities will be assessed without blood tests.

The blood samples will be tested in the research lab. Then investigators shall compare the clinical findings with the laboratory findings, and see if any of the markers found reflect the injury severity or predict the recovery.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of traumatic or non-traumatic Spinal cord injury, Guillain-barre syndrome or Stroke
* No more than 3 months after injury or disease onset
* Condition severe enough to necessitate hospital/day care unit
* Signed the informed consent form

Exclusion Criteria:

* Psychiatric or cognitive situations that may interfere with the trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients attmited for neuro-rehabilitation with spinal cord injury, stroke or Guillain-Barre syndrome
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2012-01

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel